CLINICAL TRIAL: NCT06852508
Title: TwySHE - An Mhealth Peer-navigator Intervention to Increase PrEP and Contraceptive Use Among Sexually Active Female University Students in Zambia: Study Protocol of a Hybrid Effectiveness-implementation Randomized Controlled Trial
Brief Title: TwySHE - An Mhealth Peer-navigator Intervention to Increase PrEP and Contraceptive Use
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of Zambia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 22-1151
Record Dates: First submitted 2025-02-24; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Hiv; Contraception Behavior
Keywords: HIV prevention; Modern contraception; Pre-exposure prophylaxis; PrEP
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Contraception Behavior

STUDY DESIGN:
Intervention Model Description: 1:1 individual-randomized, open-label single-site hybrid type 1 effectiveness-implementation trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TwySHE mhealth peer navigator intervention (Experimental): Trained peer navigators will promote PrEP and contraception uptake/persistence among participants by communicating with them in-person or over mobile devices twice per month for 6 months. The first visit (in-person) is focused on building rapport and a trusting relationship with the participant. During the second visit (in-person) and subsequent sessions (in-person or mobile communication), the peer navigators will focus on encouraging, supporting, and helping build the skills of their participants to address their HIV/SRH needs, provide referrals and linkage to available services, and follow up to ensure participants access those services. Subsequent visits will be conducted as needed, depending on the participant.
  Interventions: Behavioral: TwySHE
- Control (No Intervention): Participants will receive a referral list for local HIV/SRH services and informed of the longitudinal data collection process through 12 months.

INTERVENTIONS:
Behavioral: TwySHE — Interpersonal support from trained peers to access and use PrEP and contraception.
  Other Names: mhealth peer navigator intervention
  Arms: TwySHE mhealth peer navigator intervention

SUMMARY:
The goal of this clinical trial is to learn if the TwySHE intervention can increase the use of HIV prevention in at-risk female university students aged 18-24 in Zambia. The main question it aims to answer is:

• Can a mhealth peer navigator intervention effectively promote HIV pre-exposure prophylaxis PrEP use among high-risk female students in Zambia?

Researchers will compare the mhealth peer navigator intervention to treatment as usual to see if there are effects on female student's use and continuation of PrEP for HIV prevention.

Participants in the intervention will be paired with a trained peer navigator who will offer education, social support, and help navigating the health systems to access PrEP and other sexual and reproductive health services.

All participants in both arms will complete surveys at baseline, 6 months, and 12 months to evaluate health behaviors.

DETAILED DESCRIPTION:
We are conducting a 1:1 individual-randomized, open-label single-site hybrid type 1 effectiveness-implementation trial to determine the effectiveness the TwySHE intervention in Lusaka, Zambia. We will follow all participants for 12 months with regular data collection. All intervention activities will end at 6 months (primary endpoint window), but we will continue to follow and survey participants in both study arms at 12 months to determine long-term post-intervention effectiveness. PrEP and contraception uptake and persistence will be objectively verified using a study medical visit card filled out and signed by health providers. We will also collect and assess behavioral mechanisms hypothesized to be on the casual pathway, including participant knowledge regarding HIV and unintended pregnancy prevention, health beliefs (perceived risk of HIV or unintended pregnancy), perceived social support to access and adhere to HIV/unintended pregnancy prevention methods, stigma, behavioral intention to use PrEP and contraception, and self-efficacy to use PrEP and contraception. Lastly, we will conduct exit interviews with peer-navigators and a sub-sample of participants to explore the implementation outcomes of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Aged 18 to 24 years
* Current university student
* Not diagnosed with HIV
* Self-report of 3 more HIV risk factors

Exclusion Criteria:

* Male
* Less than 18 years of age
* Greater than 24 years of age
* Diagnosed with HIV
* Less than 3 self-reported HIV risk behaviors
* Not a university student

Ages: 18 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 324 (Estimated)
Dates: Start 2025-02-18 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
PrEP uptake | 6 months
  Self-reported use of PrEP products verified through health clinic documentation

SECONDARY OUTCOMES:
Contraception uptake | 6 months
  Self-reported use of PrEP products verified through health clinic documentation

OTHER OUTCOMES:
PrEP persistence | 12 months
  Self-reported continued use of PrEP if initiated verified through health clinic documentation
Contraception persistence | 12 months
  Self-reported continued use of PrEP if initiated verified through health clinic documentation

CONTACTS AND LOCATIONS:
Overall Officials: Karen M Hampanda, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Zambia, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results after deidentification
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After publication
Access Criteria: Researchers who provide a methodologically sound proposal and sign a data use agreement